CLINICAL TRIAL: NCT04764422
Title: A Phase 1/2 Randomized, Placebo-controlled, Observer-blind Trial to Assess the Safety and Immunogenicity of NDV-HXP-S Vaccine in Thailand
Brief Title: Assess the Safety and Immunogenicity of NDV-HXP-S Vaccine in Thailand
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: The Government Pharmaceutical Organization (Other Government)
Responsible Party: Principal Investigator, Punnee Pitisuttithum, Professor, Mahidol University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: GPO NDV-HXP-S
Record Dates: First submitted 2021-02-08; First posted 2021-02-21 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Covid-19; SARS Pneumonia; Pneumonia, Viral; Covid-19 Vaccine
Keywords: COVID-19; COVID-19 VACCINE; ADULT; THAILAND; GPO; The Government Pharmaceutical Organization; SAFETY; TOLERABILITY; IMMUNOGENICITY; NDV-HXP-S Vaccine; CpG1018; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Pneumonia, Viral | interventions — Saline Solution; NDV-HXP-S COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Unblinded study staff, including the site pharmacist, will be responsible for preparing study products (in accordance with the randomly determined assignment), administering the study vaccine, and handling all drug accountability procedures. These personnel will not participate in the other aspects of the clinical trial, to help ensure the integrity of the blind at the site. Unblinded staff will retrieve a subject's randomization assignment after being informed by the PI or designee that a subject is eligible for randomization. They will prepare the 0.5 ml dose of study product based on the subject's randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator): 0.9% Normal Saline for injection
  Interventions: Biological: Normal Saline
- NDV-HXP-S 1 µg (Active Comparator): 35 subjects age 18-59 will receive NDV-HXP-S 1 µg study vacine administered 0.5 mL IM
  Interventions: Biological: NDV-HXP-S vaccine
- NDV-HXP-S 3 µg (Active Comparator): 35 subjects age 18-59 will receive NDV-HXP-S 3 µg study vacine administered 0.5 mL IM
  Interventions: Biological: NDV-HXP-S vaccine
- NDV-HXP-S 10 µg (Active Comparator): 35 subjects age 18-59 will receive NDV-HXP-S 10 µg study vacine administered 0.5 mL IM
  Interventions: Biological: NDV-HXP-S vaccine
- NDV-HXP-S 1 µg + CpG1018 1.5 mg (Active Comparator): 35 subjects age 18-59 will receive NDV-HXP-S 1 µg + CpG1018 1.5 mg study vacine administered 0.5 mL IM
  Interventions: Biological: NDV-HXP-S vaccine
- NDV-HXP-S 3 µg + CpG1018 1.5 mg (Active Comparator): 35 subjects age 18-59 will receive NDV-HXP-S 3 µg + CpG1018 1.5 mg study vacine administered 0.5 mL IM
  Interventions: Biological: NDV-HXP-S vaccine

INTERVENTIONS:
Biological: Normal Saline — 0.9% normal saline for injection
  Arms: Placebo
Biological: NDV-HXP-S vaccine — Vaccine NDV-HXP-S, manufactured by GPO with or without adjuvant CpG1018.
  Arms: NDV-HXP-S 1 µg; NDV-HXP-S 1 µg + CpG1018 1.5 mg; NDV-HXP-S 10 µg; NDV-HXP-S 3 µg; NDV-HXP-S 3 µg + CpG1018 1.5 mg

SUMMARY:
This study will be conducted in 2 phases. Phase 1 designed to evaluate safety, tolerability and immunogenicity COVID-19 vaccine (NDV-HXP-S) administered at different doses levels (1, 3, and 10 µg) without adjuvant, and at two different dose levels (1 and 3 µg) with the adjuvant CpG 1018 among healthy adults, (age 18-59 years) (210 subjects). Subjects will receive 2 doses of assigned investigational product (IP) on D1 and D29 (V1 and V3), and be assessed in clinic for safety and reactogenicity at 7 days after each vaccination (day 1 as day vaccination). An interim analysis of Phase 1 data will be conducted as the basis for decisions about advancement to Phase 2 of the study and about treatment group down selection. Phase 2 (250 subjects) will include approximately one-third subjects with age 60-75 years.

DETAILED DESCRIPTION:
This study (GPO NDV-HXP-S) will be conducted in 2 phases. Phase 1 will evaluate the safety, tolerability and immunogenicity COVID-19 vaccine (NDV-HXP-S) administered at different doses levels (1, 3, and 10 µg) without adjuvant, and at two different dose levels (1 and 3 µg) with the adjuvant CpG 1018 among healthy adults, (age 18-59 years, 210 subjects). NDV-HXP-S or placebo (0.9% normal saline for injection) will administer IM according to a repeat vaccination schedule (given 28 days apart). In addition, as exploratory objectives, a total of 36 subjects will be randomly selected (1:1:1 ratio) from placebo and two high-dose groups i.e., NDV-HXP-S 10 µg and NDV-HXP-S 3 µg + CpG 1018, to provide additional blood at V1, V5 and V7 for assessment of T-cell-mediated immunity (CMI). An interim analysis of Phase 1 data will be conducted as the basis for decisions about advancement to Phase 2 of the study and about treatment group down selection.

In the Phase 2 study, 250 subjects aged 18-75 years will be randomized (1:2:2) to placebo (0.9% normal saline for injection), or one of two selected formulations of NDV HXP S being evaluated in Phase 1 will be enrolled to Phase 2 study. Twelve subjects in each of the three Phase 2 groups (distributed among the two age strata) will be randomized to provide additional blood at V1, V5 and V7 for assessment of T-cell-mediated immunity (CMI).

Unblinding will be done as per specific SOP provided by Sponsor. The PI will be expected to provide a rationale for the necessity of unblinding, based on the expectation that knowledge of the subject's treatment assignment will have a meaningful impact on the subject's medical care in the short term. If a subject's treatment assignment is unblinded, the subject will remain in the study and continue with protocol-defined study visits and procedures, unless there is another reason for subject discontinuation.

Scheduled unblinding regarding safety concern during severe COVID-19 situation:

The elderly subjects (60-75 years) who received placebo will be unblinded and discontinued as soon as COVID-19 vaccine (AstraZeneca) become available from Sponsor. If unblinding is occurred before complete enrollment of 75 elderly subjects, the randomization assignment will be skipped in placebo arm. Therefore, no further subjects will be randomly assigned to receive placebo after unblinding.

ELIGIBILITY:
Inclusion Criteria:

Phase 1 Only:

1. Adult 18 through 59 years of age, inclusive, at screening
2. Healthy, as defined by absence of clinically significant medical condition, either acute or chronic, as determined by medical history, physical examination, screening laboratory test results, and clinical assessment of the investigator.

Phase 2 Only:

1. Adult 18 through 75 years of age, inclusive, at screening.
2. Having no clinically significant acute medical condition, and no chronic medical condition that has not been controlled within 90 days of randomization, as determined by medical history, physical examination, screening laboratory test results, and clinical assessment of the investigator.

Both Phase 1 and Phase 2:

1. Has provided written informed consent prior to performance of any study-specific procedure.
2. Has a body mass index (BMI) of 17 to 40 kg/m2, inclusive, at screening.
3. Resides in study site area and is able and willing to adhere to all protocol visits and procedures.
4. If a woman is of childbearing potential, must not be breastfeeding or be pregnant (based on a negative serum pregnancy test at screening and a negative urine pregnancy test during the 24 hours prior to receipt of the first dose of IP), must plan to avoid pregnancy for at least 28 days after the last dose of IP, and be willing to use an adequate method of contraception consistently and have a repeated pregnancy test prior to the second (last) dose of IP.

Exclusion Criteria:

Phase 1 Only:

1. A positive serologic test for SARS-CoV-2 IgG test.

Both Phase 1 and Phase 2:

1. Use of any investigational medicinal product within 90 days prior to randomization or planned use of such a product during the period of study participation.
2. History of administration of any non-study vaccine within 28 days prior to administration of study vaccine or planned vaccination during the course of study participation Note: receipt of any COVID-19 vaccine that is licensed or granted Emergency Use Authorization in Thailand during the course of study participation is not exclusionary if administered after Visit 5
3. Previous receipt of investigational vaccine for SARS or MERS, or any investigational or licensed vaccine that may have an impact on interpretation of the trial results
4. History of hypersensitivity reaction to any prior vaccination or known hypersensitivity to any component of the study vaccine
5. History of egg or chicken allergy
6. History of angioedema
7. History of anaphylaxis
8. Acute illness (moderate or severe) and/or fever (body temperature measured orally ≥38°C)
9. Any abnormal vital sign deemed clinically relevant by the PI.
10. Abnormality in screening laboratory test deemed exclusionary by the PI.
11. A positive serologic test for SARS-CoV-2 IgM test, human immunodeficiency virus (HIV 1/2 Ab), hepatitis B (HBsAg) or hepatitis C (HCV Ab)
12. History of laboratory-confirmed COVID-19 (RT-PCR positive to SAR-CoV-2)
13. History of malignancy, excluding non-melanoma skin and cervical carcinoma in situ
14. Any confirmed or suspected immunosuppressive or immunodeficient state
15. Administration of immunoglobulin or any blood product within 90 days prior to first study injection or planned administration during the study period.
16. Administration of any long-acting immune-modifying drugs (e.g., infliximab or rituximab) or the chronic administration (defined as more than 14 days) of immunosuppressants within six months prior to first study injection, or planned administration during the study period (includes systemic corticosteroids at doses equivalent to ≥ 0.5 mg/kg/day of prednisone; the use of topical steroids including inhaled and intranasal steroids is permitted).
17. History of known disturbance of coagulation or blood disorder that could cause anemia or excess bleeding. (e.g, thalassemia, coagulation factor deficiencies).
18. Recent history (within the past year) or signs of alcohol or substance abuse.
19. Any medical, psychiatric or behavior condition that in the opinion of the PI may interfere with the study objectives, pose a risk to the subject, or prevent the subject from completing the study follow-up.
20. Employee of any person employed by the Sponsor, the contract research organization (CRO), the PI, study site personnel, or site.

Note: specific exclusion criteria (e.g., ≥Grade 2 acute illness, or abnormal vital sign deemed clinically relevant by the PI) will be reassessed at both vaccination visits. Any subject who cannot be vaccinated due to an acute abnormality assessed at a vaccination visit (Visit 1 or Visit 3) may return once the acute issue has resolved, if deemed appropriate by the PI. A minimum of 48 hours must have passed after a documented fever before a subject can be vaccinated. This safety requirement will not be deemed a protocol deviation should the visit fall outside the vaccination window; however, it will be encouraged to maintain the vaccination window whenever possible in these situations. Clinical laboratory test results and vital signs used to determine subject eligibility will be those obtained at screening. These tests may be repeated once if deemed appropriate by the investigator and determined to be due to a transient condition that has resolved. In addition, a test may also be repeated for test results determined to be spurious by the investigator (e.g., following improper specimen collection). The last measurement will be taken as the baseline for purposes of analysis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Frequency of solicited reportable local adverse event after first vaccination | Day 1 up to Day 7 after first vaccination
  Frequency of solicited reportable local adverse events (pain or tenderness, erythema, swelling or induration) of first vaccination
Frequency of solicited reportable local adverse event after second vaccination | Day 1 up to Day 7 after second vaccination
  Frequency of solicited reportable local adverse events (pain or tenderness, erythema, swelling or induration) of second vaccination
Frequency of solicited reportable systemic adverse event after first vaccination | Day 1 up to Day 7 after first vaccination
  Frequency of solicited reportable systemic adverse events (fever, headache,fatigue or malaise, myalgia, arthralgia,nausea or vomitting) of first vaccination
Frequency of solicited reportable systemic adverse event after second vaccination | Day 1 up to Day 7 after second vaccination
  Frequency of solicited reportable systemic adverse events (fever, headache,fatigue or malaise, myalgia, arthralgia,nausea or vomitting) of second vaccination
Measurement of hemoglobin changed from baseline at 7 days after first and second vaccination | Day 8, Day 36
  Measurement of hemoglobin (g/dl) changed from baseline at 7 days after first and second vaccination
Measurement of white blood cells changed from baseline at 7 days after first and second vaccination | Day 8, Day 36
  Measurement of white blood cells (10^3 cells/ul) changed from baseline at 7 days after first and second vaccination
Measurement of platelet count changed from baseline at 7 days after first and second vaccination | Day 8, Day 36
  Measurement of platelet count (10^3 cells/ul) changed from baseline at 7 days after first and second vaccination
Measurement of creatinine changed from baseline at 7 days after first and second vaccination | Day 8, Day 36
  Measurement of creatinine (mg/dl) changed from baseline at 7 days after first and second vaccination
Measurement of AST changed from baseline at 7 days after first and second vaccination | Day 8, Day 36
  Measurement of AST (U/L) changed from baseline at 7 days after first and second vaccination
Measurement of ALT change from baseline at 7 days after first and second vaccination | Day 8, Day 36
  Measurement of ALT (U/L) change from baseline at 7 days after first and second vaccination
Measurement of total bilirubin changed from baseline at 7 days after first and second vaccination | Day 8, Day 36
  Measurement of total bilirubin (mg/dl) change from baseline at 7 days after first and second vaccination
Frequency of all unsolicited AEs | Day 1 up to Day 56
  Frequency of all unsolicited AEs
Frequency of SAEs | Day 1 up to Day 365
  Frequency of SAEs throughout the entire study period
Frequency of medically-attended adverse event (MAAEs) | Day 1 up to Day 365
  Frequency of medically-attended adverse event (MAAEs) throughout the entire study period
Frequency of AESI | Day 1 up to Day 365
  Frequency of AESI throughout the entire study period, including AESI relevant to COVID-19, and potential immune-mediated medical conditions (PIMMC) presented as number and percentage

SECONDARY OUTCOMES:
GMT Neutralizing antibody titer 50 changed from baseline after vaccination | Day 29, Day 43, Day 197, Day 365
  GMT Neutralizing antibody titer 50 changed from baseline after vaccination
GMT Neutralizing antibody titer 80 changed from baseline after vaccination | Day 29, Day 43, Day 197, Day 365
  GMT Neutralizing antibody titer 80 changed from baseline after vaccination
NT50 seroresponses changed from baseline after vaccination | Day 29, Day 43, Day 197, Day 365
  Frequency of subjects with NT50 seroresponses against SARS-CoV-2 pseudovirus as defined by (1) a ≥ 4-fold increase from baseline, and (2) a ≥ 10-fold increase from baseline after vaccination
NT80 seroresponses changed from baseline after vaccination | Day 29, Day 43, Day 197, Day 365
  Frequency of subjects with NT80 seroresponses against SARS-CoV-2 pseudovirus as defined by (1) a ≥ 4-fold increase from baseline, and (2) a ≥ 10-fold increase from baseline after vaccination
GMT Anti-S IgG after vaccination | Day 29, Day 43, Day 197, Day 365
  GMT Anti-S IgG after vaccination in subjects who are anti-S IgG seronegative at baseline
GMFR changed from baseline in anti-S IgG GMT after vaccination | Day 29, Day 43, Day 197, Day 365
  GMFR changed from baseline in anti-S IgG GMT after vaccination
Anti-S IgG Seroresponses changed from baseline after vaccination | Day 29, Day 43, Day 197, Day 365
  Frequency of subjects with seroresponses in anti-S IgG titer as defined by (1) a ≥ 4-fold increase from baseline, and (2) a ≥ 10-fold increase from baseline after vaccination

OTHER OUTCOMES:
S protein-specific T cells response changed from baseline after vaccination | Day 43, Day 197
  Frequency of S protein-specific T cells relative to baseline after vaccination
Anti-NDV HN GMT changed from baseline after vaccination | Day 29, Day 43, Day 197, Day 365
  Anti-NDV HN GMT changed from baseline after vaccination
Anti-NDV HN IgG GMT changed from baseline after vaccination | Day 29, Day 43, Day 197, Day 365
  Anti-NDV HN IgG GMT changed from baseline after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Punnee Pitisutthithum, Principal Investigator — Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University
Locations (1):
- Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
data or left over specimen will be shared for future study ONLY subject who consent allow using their data/specimens. Sharing will be done without personnel identification
Supporting Information: Study Protocol, SAP
Time Frame: 2 years after vaccine marketing
Access Criteria: as document attach when completed study in NCT clinicaltrials.gov

REFERENCES:
- [Derived] Pitisuttithum P, Luvira V, Lawpoolsri S, Muangnoicharoen S, Kamolratanakul S, Sivakorn C, Narakorn P, Surichan S, Prangpratanporn S, Puksuriwong S, Lamola S, Mercer LD, Raghunandan R, Sun W, Liu Y, Carreno JM, Scharf R, Phumratanaprapin W, Amanat F, Gagnon L, Hsieh CL, Kaweepornpoj R, Khan S, Lal M, McCroskery S, McLellan J, Mena I, Meseck M, Phonrat B, Sabmee Y, Singchareon R, Slamanig S, Suthepakul N, Tcheou J, Thantamnu N, Theerasurakarn S, Tran S, Vilasmongkolchai T, White JA, Bhardwaj N, Garcia-Sastre A, Palese P, Krammer F, Poopipatpol K, Wirachwong P, Hjorth R, Innis BL. Safety and immunogenicity of an inactivated recombinant Newcastle disease virus vaccine expressing SARS-CoV-2 spike: Interim results of a randomised, placebo-controlled, phase 1 trial. EClinicalMedicine. 2022 Mar 8;45:101323. doi: 10.1016/j.eclinm.2022.101323. eCollection 2022 Mar. PMID 35284808
- [Derived] Pitisuttithum P, Luvira V, Lawpoolsri S, Muangnoicharoen S, Kamolratanakul S, Sivakorn C, Narakorn P, Surichan S, Prangpratanporn S, Puksuriwong S, Lamola S, Mercer LD, Raghunandan R, Sun W, Liu Y, Carreno JM, Scharf R, Phumratanaprapin W, Amanat F, Gagnon L, Hsieh CL, Kaweepornpoj R, Khan S, Lal M, McCroskery S, McLellan J, Mena I, Meseck M, Phonrat B, Sabmee Y, Singchareon R, Slamanig S, Suthepakul N, Tcheou J, Thantamnu N, Theerasurakarn S, Tran S, Vilasmongkolchai T, White JA, Garcia-Sastre A, Palese P, Krammer F, Poopipatpol K, Wirachwong P, Hjorth R, Innis BL. Safety and Immunogenicity of an Inactivated Recombinant Newcastle Disease Virus Vaccine Expressing SARS-CoV-2 Spike: Interim Results of a Randomised, Placebo-Controlled, Phase 1/2 Trial. medRxiv [Preprint]. 2021 Sep 22:2021.09.17.21263758. doi: 10.1101/2021.09.17.21263758. PMID 34580673